CLINICAL TRIAL: NCT07245797
Title: the Efficacy and Safety of Neoadjuvant Therapy With Inavolisib Plus Pertuzumab and Trastuzumab as Subcutaneous (PH-FDC SC) and 3-week Cycle Nab-paclitaxel for PIK3CA-mutated, HER2+, eBC
Brief Title: A Phase II, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of Neoadjuvant Therapy With Inavolisib Plus Pertuzumab and Trastuzumab as Subcutaneous (PH-FDC SC) and 3-week Cycle Nab-paclitaxel for PIK3CA-mutated, HER2+, eBC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhimin Shao (Other)
Responsible Party: Sponsor-Investigator, Zhimin Shao, Director, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2509329-18
Record Dates: First submitted 2025-09-30; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; 130-nm albumin-bound paclitaxel; inavolisib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fixed-dose combination of pertuzumab and trastuzumab，and nab-paclitaxel with inavolisib. (Experimental)
  Interventions: Drug: fixed-dose combination of pertuzumab and trastuzumab as subcutaneousformulation q3w and nab-paclitaxel in 3-week cycle for total 6 cycles with inavolisib (6 cycles) or without inavolisib.
- fixed-dose combination of pertuzumab and trastuzumab，and nab-paclitaxel. (Active Comparator)
  Interventions: Drug: fixed-dose combination of pertuzumab and trastuzumab as subcutaneousformulation q3w and nab-paclitaxel in 3-week cycle for total 6 cycles with inavolisib (6 cycles) or without inavolisib.

INTERVENTIONS:
Drug: fixed-dose combination of pertuzumab and trastuzumab as subcutaneousformulation q3w and nab-paclitaxel in 3-week cycle for total 6 cycles with inavolisib (6 cycles) or without inavolisib. — fixed-dose combination of pertuzumab and trastuzumab as subcutaneousformulation q3w and nab-paclitaxel in 3-week cycle for total 6 cycles with inavolisib (6 cycles) or without inavolisib.

SUMMARY:
The study consists of a screening period of 28 days, a treatment period. Local or central testing of PIK3CA mutation in blood or tumor tissue must be performed using an approved polymerase chain reaction (PCR)-based or next generation sequencing (NGS) assay at a clinical laboratory. Patients with confirmed eligibility criteria and PIK3CA mutant breast cancer will be randomized in a 1:1 ratio to receive:

Neoadjuvant treatment with dual anti-HER2 blockade consisting of ready-to-use fixed-dose combination of pertuzumab and trastuzumab as subcutaneous (PH-FDC SC) formulation q3w and nab-paclitaxel (125 mg/m2 on days 1, 8, and 15) in 3-week cycle for total 6 cycles

* with inavolisib (6 cycles) or
* without inavolisib. In both study arms, treatment will be given until surgery/core-biopsy, disease progression, unacceptable toxicity, or withdrawal of consent of the patient.

All patients will undergo surgery or biopsy after completing study therapy to assess pCR rate.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for study participation only if they comply with the following criteria:

1. Written informed consent for all study procedures according to local regulatory requirements prior to beginning specific protocol procedures.
2. Untreated, unilateral primary carcinoma of the breast, confirmed histologically by core biopsy. Fine-needle aspiration alone is not sufficient. Incisional biopsy is not allowed.
3. Tumor lesion in the breast must be measurable in two dimensions, preferably by sonography.
4. Patients must be in the following stages of disease:

   •cT1b - cT3 regardless of nodal status. In patients with multifocal or multicentric breast cancer the largest lesion (target lesion) should be measured.
5. HER2+ disease with confirmed ER-status, PR-status, HER2-status, PIK3CA mutation (tumor), Ki-67 value on core biopsy (target lesion). HER2-positive is defined according to current ASCO/CAP Guidelines. PIK3CA needs to be tested at the local site.
6. Age ≥ 18 years, female and male.
7. ECOG Performance status 0-1.
8. Normal cardiac function must be confirmed by ECG and cardiac ultrasound (LVEF or shortening fraction) within 3 months prior to randomization. Results for LVEF must be above 55%.
9. Laboratory requirements:

   Hematology
   * Absolute neutrophil count (ANC) ≥ 1.5/ nL
   * Platelets ≥ 100/ nL and
   * Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L) Hepatic function
   * Total bilirubin < ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN
   * AST and ALT ≤ 1.5x ULN and
   * Alkaline phosphatase ≤ 2.5x ULN

   Glucose Metabolism:
   * Glycosylated hemoglobin (HbA1c) < 6.5%
   * Fasting plasma glucose (FPG) < 126 mg/dL (7.0 mmol/L)
10. Staging work-up according to country guidelines prior to randomization including:

    ● Bilateral mammography and/or breast MRI in combination with a breast ultrasound. Exception: In men where MRI is medically not indicated breast ultrasound is sufficient.
11. Patients must be willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
12. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs, as defined below: Women must remain abstinent or use non-hormonal contraceptive methods with a failure rate of 1% per year during the treatment period and for at least 60 days after the final dose of study treatment. Based on local prescribing information for fulvestrant, patients may be advised to use an effective means of contraception for up to 2 years after the final dose of fulvestrant. Women must refrain from donating eggs during this same period.
13. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state ( 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations. Examples of non-hormonal contraceptive methods with a failure rate of 1% per year include bilateral tubal ligation, male sterilization, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. If required per local guidelines or regulations, locally recognized acceptable methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

Exclusion Criteria:

Patients will be ineligible for study participation if they comply with the following criteria:

1. Patients with HER2-negative breast cancer.
2. Inflammatory breast cancer.
3. Patients with definitive clinical or radiologic evidence of Stage IV cancer or bilateral breast cancer or invasive breast cancer.
4. Excisional biopsy or lumpectomy and/or axillary lymph node dissection and/or sentinel lymph node biopsy performed prior to study entry (biopsy of clinical involved LN is warranted).
5. Prior chemotherapy or endocrine therapy or radiation therapy prior to study entry with the following exceptions:

   •If medically indicated, initiation of hormonal replacement therapy (HRT) up to 28 days prior to randomization and use of established fertility preservation methods (including Gn) in young patients interested in subsequent pregnancies is allowed.
6. Patients with a history of any treated malignancy and/or ongoing oncological treatment are ineligible, excluding cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin. This also applies to patients who are at high risk that oncological treatment is indicated during study therapy.
7. Known hypersensitivity reaction to one of the compounds or substances, and/or murine proteins, and/or recombinant human hyaluronidase used in this protocol.
8. Patients with an established diagnosis of diabetes mellitus type I or uncontrolled type II based on FPG and HbA1c (refer to Inclusion Criteria No.10）.
9. Type II diabetes requiring ongoing systemic treatment at the time of study entry or any history of Type 1 diabetes.
10. Patients who are known HIV infection if any of the following apply: The CD4+ count is less than 350 cells/uL or there has been an opportunistic infection within the 12 months prior to the start of study treatment. Patients who are known to have HIV infection receiving immunosuppressive therapies and there is a potential DDI with any of the study treatments.
11. Clinically significant and active liver disease, for example, sclerosing cholangitis, active viral hepatitis B or C infection, or autoimmune hepatic disorders.
12. Patients with inflammatory bowel disease, such as Crohn's disease or ulcerative colitis, and active bowel inflammation (e.g., diverticulitis).
13. Patients with any concurrent ocular or intraocular condition, excluding baseline cataracts, require medical or surgical intervention during the study period to prevent or treat vision loss. In addition, patients with active uveitis or vitritis, history of uveitis, or active infectious process in the eye.
14. Patients with Previously or currently documented pneumonitis/interstitial lung disease, except if the investigator determines that it is non-active and does not require corticosteroid treatment.
15. Known or suspected congestive heart failure (>NYHA I) and / or coronary heart disease, angina pectoris requiring antianginal medication, previous history of myocardial infarction, evidence of transmural infarction on ECG, uncontrolled or poorly controlled arterial hypertension (i.e. BP>160/90 mm Hg under treatment with three antihypertensive drugs), rhythm abnormalities requiring permanent treatment, clinically significant valvular heart disease.
16. Damaged skin at planned site of subcutaneous (SC) injections (thigh).
17. Patients who may have had a recent episode of thromboembolism and are still trying to optimize the anticoagulation dose and/or have not normalized their INR.
18. Concurrent treatment with:

    * Systemic chronic corticosteroids < 2 weeks prior to starting study treatment or has not recovered from side effects of such treatment The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops, or local injections (e.g., intra-articular). Except if chronic corticosteroids initiated >6 months prior to study entry and at low dose (10 mg or less methylprednisolone or equivalent).
    * Sex hormones. Prior treatment must be stopped before randomization.
    * Other experimental drugs or any other anti-cancer therapy.
19. Participation in another clinical trial with any investigational drugs, not marketed drug within 30 days prior to study entry.
20. Female patients: pregnancy or lactation at the time of randomization.
21. History of significant neurological or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent.
22. Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
23. Pregnant, lactating, or breastfeeding, or intending to become pregnant during the study or within 60 days after the final dose of study treatment. Women of childbearing potential (including those who have had a tubal ligation) must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-02-23 (Estimated)

PRIMARY OUTCOMES:
pCR（ypT0/is ypN0） | 6months
  pCR (ypT0/is ypN0) is defined as the absence of microscopically residual invasive tumor cells in all resected specimens from the breast and axilla. Pathological response will be comprehensively evaluated based on all surgically resected breast and lymph node tissues. Biopsy alone is insufficient to confirm pCR; patients with no residual tumor in the biopsy should undergo surgery (otherwise, they are considered not to have achieved pCR, as are all patients for whom pCR cannot be confirmed). Patients who receive additional treatment after biopsy or without prior biopsy, regardless of the subsequent neoadjuvant treatment response, are considered not to have achieved pCR. Before surgical evaluation to confirm pCR, additional neoadjuvant treatment should be avoided after the completion of the study treatment.

SECONDARY OUTCOMES:
ypT0 | 6months
  ypN0 is defined as the absence of microscopic evidence of residual invasive or non-invasive viable tumor cells in all resected specimens from the breast and axilla; ypT0 ypN0/+ is defined as the absence of microscopic evidence of residual invasive or non-invasive viable tumor cells in all resected specimens from the breast; ypT0/Tis ypN0/+ is defined as the absence of microscopic evidence of residual invasive viable tumor cells in all resected specimens from the breast.
ORR | 6months
  Objective Response Rate (ORR) is defined as the proportion of patients who achieve a best overall response of Complete Response (CR) or Partial Response (PR) during neoadjuvant therapy, as assessed by the investigator according to RECIST v1.1 criteria.
safety | 6 months
  The severity of adverse events was determined using the NCI-CTC AE 5.0 standard. During the trial, the adverse event record form should be filled in truthfully, including the time of occurrence, severity, relevance to the study treatment, duration, measures taken, and outcome of the adverse event.

OTHER OUTCOMES:
Exploratory end points | 1 year
  Explore novel biomarkers based on collected samples of tumor tissue, adjacent normal tissue, and blood from subjects, and investigate the association between biomarkers and the disease status or treatment response of the subjects.